CLINICAL TRIAL: NCT00280410
Title: Multicenter, Randomized, Open-Label Study Investigating The Superiority Of The Contrast Enhancement Effect Of E7337 On Tumor Like Lesion In The Dynamic CT Of The Liver Of Patients With Tumor Like Lesions In The Liver
Brief Title: Study Investigating the Effect of E7337 on Tumor Like Lesions in Computed Tomography (CT) of the Liver
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: Eisai Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: E7337-J081-151
Record Dates: First submitted 2006-01-20; First posted 2006-01-23 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2010-01

CONDITIONS: Lesions of the Liver

INTERVENTIONS:
Drug: E7337

SUMMARY:
This is a multicenter, randomized, open-label study to investigate the superiority of the contrast enhancement effect of E7337 on tumor-like lesions in the Dynamic CT of the liver.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a tumorous lesion in the liver observed in diagnostic imaging such as ultrasonography, etc., conducted between 1 and 35 days before administration of the investigational agent, who are scheduled to undergo a dynamic CT examination.
2. Patients between 20 and 80 years old at the time informed consent is obtained.
3. Patients weighing >= 55.6 and < 105.0 kg at the time consent is obtained and when the investigational agent is administered.

Exclusion Criteria:Issues affecting the safety evaluation of the investigational agent:

1. Patients who will have undergone or are scheduled to undergo an examination using another contrast agent from 7 days before administration of the investigational agent up to the time follow-up examinations are performed on day 8 after administration.
2. Patients for whom there is a strong possibility that a follow-up period, which extends up until examinations are performed on day 8 after administration, would not be possible, (i.e., when it will not be possible to evaluate delayed adverse drug reactions).
3. Patients who have undergone or are scheduled to undergo surgical treatment or a therapy such as percutaneous ethanol injection therapy, percutaneous microwave coagulation therapy, radiofrequency ablation, or transcatheter arterial embolization, etc., from the time diagnostic imaging such as abdominal ultrasonography is performed up until follow-up examinations are conducted on day 8 after administration.
4. Patients who are unable to discontinue taking analgesics during the period from the morning when the investigational agent is administered until CT examinations are completed.
5. Patients who cannot stop taking biguanide antidiabetic drugs, such as metformin hydrochloride and buformin hydrochloride, for three days after study agent administration (including administration day).
6. Patients who are currently participating in another clinical study.
7. Patients who participated in another clinical study within the 6 months prior to providing informed consent to participate in this study.

General concerns relating to the safety of the subject:

1. Patients in the acute stage of illness with unstable symptoms, or patients in a life-threatening condition (when it is expected that emergency treatment may be required between the time of registration and the conclusion of the follow-up period, or when the patient is not expected to survive for 3 months following administration of the investigational agent, etc.)
2. Patients with a history of hypersensitivity to iodine or iodinated contrast agents.
3. Patients with serious thyroid disease (goiter, hyperthyroidism, etc.)
4. Patients with serious cardiopathy (New York Heart Association [NYHA] functional class IV heart failure, shock, cyanosis, peripheral circulatory insufficiency, ventricular tachycardia, ventricular fibrillation, or complete atrioventricular block)
5. Patients with serious hepatopathy [symptoms of liver failure (fulminant hepatitis) such as a disturbance of consciousness corresponding to grade 3 in the Criteria for Grading Adverse Drug Reactions of Medicinal Products.]
6. Patients with moderate serious nephropathy (acute kidney failure, chronic kidney failure, hydronephrosis, nephrotic syndrome, or uremia with serum creatinine levels of 2.0 mg/dL or more, corresponding to grade 2 or above in the Criteria for Grading Adverse Drug Reactions of Medicinal Products.)
7. Patients with bronchial asthma
8. Patients with acute pancreatitis
9. Patients with macroglobulinemia
10. Patients with multiple myeloma
11. Patients with tetany
12. Patients with pheochromocytoma or who are suspected of having pheochromocytoma
13. Pregnant and potentially pregnant women, and nursing mothers
14. Patients with a history of medicine hypersensitivity
15. Patients with serious myasthenia gravis
16. Patients judged by an investigator for any other reason to be ineligible for participation as a subject in this study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192
Dates: Start 2006-02; Primary Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Contrast enhancement effect on tumor-like lesions in the liver.

SECONDARY OUTCOMES:
Contrast enhancement effect (amount of change in CT value) on the portal venous phase (portal vein, left and right lobes of the liver parenchyma). Contrast enhancement effect on the arterial phase (hepatic artery).

CONTACTS AND LOCATIONS:
Overall Officials: Koichi Tazawa, Study Director — Eisai Company Lmited
Locations (14):
- Japan (14):
  - Fukuoka, Fukuoka
  - Fukushima, Fukushima
  - Sapporo, Hokkaido
  - Kobe, Hyōgo
  - Kanazawa, Ishikawa-ken
  - Isehara, Kanagawa
  - Kumamoto, Kumamoto
  - Kashihara, Nara
  - Okayama, Okayama-ken
  - Sayama, Osaka
  - Suita, Osaka
  - Minato-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Shinjuku-ku, Tokyo